CLINICAL TRIAL: NCT06855784
Title: Time-Restricted Eating to Improve Body Composition and Symptoms in Menopause and HOrmone-sensitive Breast Cancers (TREMHO) - An Open-label Randomized Controlled Trial
Brief Title: Time-Restricted Eating in Menopause and HOrmone-sensitive Breast Cancers (TREMHO)
Acronym: TREMHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Tinh-Hai Collet, MD, Assistant Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01257
Record Dates: First submitted 2025-02-15; First posted 2025-03-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Menopause; Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Trehalase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Time-Restricted Eating 16h/8h
- Active Control (Active Comparator)
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Time-Restricted Eating 16h/8h — Participants will be advised to eat only during a self-selected window of 8 hours over the 24-hour cycle, with a 1-hour allowance according to their daily routine.
  Other Names: TRE 16h/8h
  Arms: Time-Restricted Eating
Behavioral: Active Control — Participants will be advised to eat 2 to 3 meals every day according to their eating habits and social activities
  Arms: Active Control

SUMMARY:
This study is aimed at women currently going through menopause, either as part of the natural process (physiological menopause), or following hormonal treatment for breast cancer. There are several ways of slowing the weight gain frequently encountered in this situation, reducing the intensity of menopause-related symptoms and improving quality of life in this context.

In this trial, the investigators examine the efficacy and possible adverse effects of intermittent fasting compared with a control intervention. Participation lasts 14 weeks, with an optional 12-month follow-up. Study participants are randomly assigned to either the intervention group or the control group. In the intervention group, study participants fast for 16 hours per day and eat over a period of 8 hours (intermittent fasting often called time-restricted eating [TRE] 16h/8h). In the control group, the usual eating pattern is continued for 12 weeks.

The main objective of the study is to evaluate the efficacy of TRE in terms of weight and fat loss, improvement in metabolic profile, menopausal symptoms and bone health. In addition, the study team closely monitors any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed physiological menopause without current anti-cancer treatment (group A), or women with menopausal symptoms in the context of aromatase inhibitors used as adjuvant therapy for hormone-sensitive non-metastatic breast cancers regardless of physiological menopause before the cancer diagnosis (group B)
* Age 40-65 years
* Body mass index 25-40 kg/m2
* Stable weight (± 2 kg) over the previous month
* Eating window ≥ 12 hours (self-reported and measured during the run-in phase)
* Able to give informed consent and follow the study procedures for the entire duration
* Confident use of a smartphone and able to take regular pictures of food/drinks

Exclusion Criteria:

* On a hypocaloric restrictive diet, intermittent fasting or in a weight management program over the previous month
* Previous bariatric surgery or planned during the study
* Active eating disorder(s) or major mental illness at inclusion
* Psychoactive treatment with recent or planned changes of drug compound or dosage
* Treatments affecting body weight (e.g. glucocorticoids, GLP-1 receptor analogues)
* Diabetes with hypoglycemic drug(s) will be excluded, however those with prediabetes (as defined by the American Diabetes Association) or diabetes with no risk of hypoglycemia (i.e. treated with non-hypoglycemic drugs or without medication) will be included
* Active metabolic bone diseases (e.g. Paget disease, osteomalacia), however women with osteoporosis will be included
* Shift work comprising night shifts (working between 11pm and 6am) over the previous 2 weeks or planned during the study
* Travel/trip to a different time zone (≥ 2-hour time difference) over the previous 2 weeks or planned during the study
* Enrolled in another interventional clinical trial (medication, surgery, medical device) over the previous 2 weeks or planned during the study

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | From randomization visit to close-out visit (12 weeks)
  Measured (in Kg) in light clothing using a calibrated medical-grade scale
Changes in body fat mass | From randomization visit to close-out visit (12 weeks)
  Measured (in Kg) by dual-energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Changes in menopause / climacteric symptoms | From randomization visit to close-out visit (12 weeks)
  Assessed by questionnaire
Changes in bone mineral density | From randomization visit to close-out visit (12 weeks)
  Measured (in g/cm3) by dual-energy x-ray absorptiometry (DXA)
Changes in bone turnover marker CTX | From randomization visit to close-out visit (12 weeks)
  C-telopeptide cross-linked type 1 collagen (CTX) measured (in ng/L) by clinical chemistry
Changes in bone turnover marker P1NP | From randomization visit to close-out visit (12 weeks)
  Procollagen type 1 N-terminal propeptide (P1NP) measured (in μg/L) by clinical chemistry
Changes in joint pain | From randomization visit to close-out visit (12 weeks)
  Joint pain assessed by questionnaire (0 = absent to 7 = Extremely bothered)
Changes in body mass index (BMI) | From randomization visit to close-out visit (12 weeks)
  Expressed in percent of baseline value (body mass index = weight in Kg divided by the height in meters squared, unit Kg/m2)
Changes in waist circumference | From randomization visit to close-out visit (12 weeks)
  Measured (in cm) with a measuring tape, following the WHO 2008 Expert Report
Changes in hip circumference | From randomization visit to close-out visit (12 weeks)
  Measured (in cm) with a measuring tape, following the WHO 2008 Expert Report
Changes in systolic and diastolic blood pressure | From randomization visit to close-out visit (12 weeks)
  Measured (in mmHg) with an arm cuff in the sitting position
Changes in fasting plasma glucose | From randomization visit to close-out visit (12 weeks)
  Measured (in mmol/L) by clinical chemistry
Changes in lipid profile | From randomization visit to close-out visit (12 weeks)
  Total cholesterol, LDL cholesterol, triglycerides and HDL cholesterol concentrations measured (in mmol/L) by clinical chemistry
Changes in lean body mass | From randomization visit to close-out visit (12 weeks)
  Measured (in Kg) by dual-energy x-ray absorptiometry (DXA)
Changes in body composition | From randomization visit to close-out visit (12 weeks)
  Fat mass and fat-free mass (in Kg) measured by bioelectrical impedance analysis (BIA)
Changes in muscle function | From randomization visit to close-out visit (12 weeks)
  Measured (in Kg) by handgrip strength
Changes in glucose excursion | From randomization visit to close-out visit (12 weeks)
  Measured by continuous glucose monitoring
Changes in metabolomic profile | From randomization visit to close-out visit (12 weeks)
  Measured by high-throughput mass spectrometry metabolomics
Changes in physical activity | From randomization visit to close-out visit (12 weeks)
  Measured by actigraphy (in activity counts, CamNTech proprietary algorithm) and by the International Physical Activity Questionnaire (IPAQ, aggregated in MET-minutes/week)
Changes in sleep/wake cycles | From randomization visit to close-out visit (12 weeks)
  Measured by actigraphy assessed as time of sleep onset and wake-up in 24-hour cycle
Changes in sleep duration | From randomization visit to close-out visit (12 weeks)
  Measured by actigraphy
Changes in body temperature | From randomization visit to close-out visit (12 weeks)
  Measured by body temperature wearable device
Changes in sleep quality | From randomization visit to close-out visit (12 weeks)
  Assessed by the Pittsburgh Sleep Quality Index [PSQI, minimum score = 0 (better); maximum score = 21 (worse)]
Changes in eating duration | From randomization visit to close-out visit (12 weeks)
  Duration from the first to last caloric intake over 24-hour cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided